CLINICAL TRIAL: NCT01497327
Title: An Open-Label Study to Characterize the Pharmacokinetics and Pharmacodynamics of Multiple Oral Doses of PSI-7977 or PSI-352938 in HCV-infected Subjects With Varying Degrees of Hepatic Impairment
Brief Title: Open-Label Hepatic Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2938-0515
Record Dates: First submitted 2011-11-30; First posted 2011-12-22 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Hepatitis C
Keywords: HEPATITIS C, CHRONIC; HCV; hepatic impairment
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — PSI 352938; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- PSI-352938 Group A (Experimental): Mild (Child-Pugh Class A; 5-6) hepatic impairment
  Interventions: Drug: PSI-352938
- PSI-352938 Group B (Experimental): Moderate (Child-Pugh Class B; 7-9) hepatic impairment
  Interventions: Drug: PSI-352938
- PSI-352938 Group C (Experimental): Severe (Child-Pugh Class C; 10-15) hepatic impairment
  Interventions: Drug: PSI-352938
- PSI-7977 Group A (Experimental): Mild (Child-Pugh Class A; 5-6) hepatic impairment
  Interventions: Drug: PSI-7977
- PSI-7977 Group B (Experimental): Moderate (Child-Pugh Class B; 7-9) hepatic impairment
  Interventions: Drug: PSI-7977
- PSI-7977 Group C (Experimental): Severe (Child-Pugh Class C; 10-15) hepatic impairment
  Interventions: Drug: PSI-7977

INTERVENTIONS:
Drug: PSI-352938 — PSI-352938 300mg once daily (QD) for seven days
  Arms: PSI-352938 Group A; PSI-352938 Group B; PSI-352938 Group C
Drug: PSI-7977 — PSI-7977 400mg QD for seven days
  Arms: PSI-7977 Group A; PSI-7977 Group B; PSI-7977 Group C

SUMMARY:
This study will be conducted in Hepatitis C positive patients to determine whether the pharmacodynamic effects of PSI-7977 or PSI-352938 are similar to HCV-infected patients with normal hepatic function, which may allow inclusion of patients with cirrhosis and varying degrees of hepatic dysfunction in future clinical studies.

DETAILED DESCRIPTION:
This study is designed per the Food and Drug Administration (FDA) guidance for patients with impaired hepatic function to assess the influence of hepatic impairment on the PK and pharmacodynamics (PD) of PSI-7977 and PSI-352938 This study will be conducted in Hepatitis C positive patients to ascertain whether the PD effects of PSI-7977 or PSI-352938 are similar to HCV-infected patients with normal hepatic function, which may allow inclusion of patients with cirrhosis and varying degrees of hepatic dysfunction in future clinical studies. Data from subjects who participated in the P2938-0212 study (PSI-352938 MAD) will be used as the control group. These subjects were documented non-cirrhotic subjects with normal hepatic function. Hepatitis C Virus (HCV) Genotypes 1-6 will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic impaired Males or females of non-childbearing potential aged > 18 years with Chronic HCV-infection
* Naïve to all direct acting anti-viral (DAA) treatments for chronic HCV infection.
* Documented Cirrhosis

Exclusion Criteria:

* Prior PEG/RBV null responders.
* Unstable cardiac disease, recent Myocardial infarction, or family history of QTc prolongation or unexplained cardiac arrest.
* Positive test at Screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, or anti-human immunodeficiency virus (HIV) Ab.
* History of clinically significant medical condition associated with other chronic liver disease
* Any current signs or symptoms of severe hepatic encephalopathy
* History of gastric or esophageal variceal bleeding in which varices have not been adequately treated with medication and surgical procedures
* Prior placement of a portosystemic shunt
* History of hepatorenal, or hepatopulmonary syndrome.
* Active spontaneous bacterial peritonitis.
* Use of medications associated with QT prolongation within 28 days prior to dosing.
* Current Hypotension
* History of Torsades de Pointes, evidence of an active or suspected cancer, or a history of malignancy, Abnormal hematological and biochemical parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic data derived from plasma samples collected over 7 days | 28 time points over Seven Days
  To characterize the pharmacokinetics (PK) of PSI-352938 over 7 days of dosing with PSI-352938 in HCV-infected patients with varying degrees of hepatic impairment compared to historical PK data.
Pharmacokinetic comparison with historical data over 7 days of dosing with PSI-7977 | Seven Days
  To characterize the PK of PSI-7977 and metabolites over 7 days of dosing with PSI-7977 in HCV-infected patients with varying degrees of hepatic impairment compared to historical PK data.

SECONDARY OUTCOMES:
Number and severity of adverse events | Seven Days
  To assess the safety and tolerability of 7 days of dosing of PSI-352938 or PSI-7977 in HCV infected patients with varying degrees of hepatic impairment.
Viral dynamics/ changes in HCV (ribonucleic acid) RNA | Baseline through follow-up (post-Day 14)
  To evaluate the viral dynamics as measured by changes in the HCV RNA in HCV-infected patients with varying degrees of hepatic impairment after 7 days of dosing with PSI-352938 or PSI-7977.
Changes in genotypic or phenotypic measurements | Seven Days
  To assess the presence of baseline polymorphisms in viral isolates and development of viral genotypic and phenotypic changes from baseline.
Dosage adjustment in hepatically impaired patients | Seven days
  To provide dosage adjustment guidance for PSI-352938 or PSI-7977 based on the degree of hepatic impairment, if applicable.

CONTACTS AND LOCATIONS:
Locations (2):
- San Antonio, Texas, United States
- San Juan, Puerto Rico, Puerto Rico